CLINICAL TRIAL: NCT04444466
Title: A First-In-Human, Randomized, Participant-Blind, Investigator-Blind, Placebo-Controlled, Single- and Multiple-Dose, Dose-Escalating Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of UCB8600 in Healthy Participants, Atopic Participants, and Chronic Spontaneous Urticaria Participants
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of UCB8600 in Healthy Participants, Atopic Participants, and Chronic Spontaneous Urticaria Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: internal company decision; not safety related
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0086; 2019-002981-12 (EudraCT Number)
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Healthy Study Participants; Chronic Spontaneous Urticaria
Keywords: Healthy study participants; UCB8600; Phase 1; Chronic spontaneous urticaria; CSU; IgE; Atopic participants; Urticaria; UCB; Food Effect (Part D)
MeSH Terms: conditions — Chronic Urticaria; Urticaria

STUDY DESIGN:
Intervention Model Description: Cohort design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an investigator- and participant-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCB8600 (Experimental): Study participants randomized to this arm will receive various single doses and multiple doses of UCB8600 administered to various cohorts.
  Interventions: Drug: UCB8600
- Placebo (Placebo Comparator): Study participants randomized to this arm will receive various single doses and multiple doses of Placebo administered to various cohorts.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: UCB8600 — Study participants will receive UCB8600 in a pre-specified sequence during the Treatment Period.
  Arms: UCB8600
Other: Placebo — Study participants will receive Placebo in a pre-specified sequence during the Treatment Period matching UCB8600.
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess safety, tolerability and pharmacokinetics (PK) of oral UCB8600.

DETAILED DESCRIPTION:
The Study was only open for recruitment of Healthy Study Participants (Part A) prior to termination and did not enroll any patient population.

ELIGIBILITY:
Inclusion Criteria:

Applicable to Parts A-D

* Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent
* Participants who are overtly healthy (in the opinion of the investigator) as determined by medical evaluation including medical history (any chronic and acute illness), physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory screening tests at the Screening Visit
* Body weight 45 kg or greater and body mass index (BMI) within the range 19 and 30 kg/m^2 (inclusive)

Part B-specific

* Study participants must have a Screening serum immunoglobulin E (IgE) of ≥30 kU/L and ≤700 kU/L for inclusion in Cohort 1 through Cohort 4a and >700 kU/L for inclusion in Cohort 4b
* Study participants must be documented to be sensitized to at least 1 common aeroallergen confirmed by (skin prick test (SPT) at Screening)

Part C-specific

* Study participants must have a diagnosis of chronic spontaneous urticaria (CSU) diagnosed by a dermatologist, allergist or clinical immunologist and have persistent symptoms most days of the week for the last 6 weeks despite regular use of an H1 antihistamine according to the EAACI/GA²LEN/EDF/WAO guideline
* Study participants must have a documented 7-day Urticaria Assessment Score (UAS7) score of 16 or above and an 7-day Itch Severity Score (ISS7) of 8 or above at Visit 2 (Day -1, Admission)
* Study participants must have a Screening serum immunoglobulin E (IgE) of ≥30 kU/L

Exclusion Criteria:

Applicable to Parts A-D

* Participant has any (acute or chronic [including severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection]) medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Study participant has 12-lead electrocardiogram (ECG) with changes considered to be clinically significant (eg, QT interval corrected using Fridericia's formula (QTcF) >450 msec , left bundle branch block, or evidence of myocardial ischemia) at the Screening Visit or Day -1 (Admission)
* A history of additional risk factors for Torsades de pointes (TdP) (eg, heart failure, hypokalemia, family history of Long QT Syndrome)
* Study participant has a history of atopy, allergic rhinitis, urticaria, angioedema, asthma, food allergies, or anaphylaxis
* Study participant has a known hypersensitivity to any components of the study medication or comparative drugs as stated in this protocol
* Study participant has a history of drug allergy or other allergy that, in the opinion of the investigator or UCB Study Physician, contraindicates his/her participation
* Study participants with evidence of helminthic parasitic infection as evidenced by stools being positive for a pathogenic organism according to local guidelines. All participants will be screened at Screening. If stool testing is positive for pathogenic organism, the participants will not enter Treatment Period and will not be allowed to rescreen
* Study participant has received prescription or nonprescription medicines (including over-the-counter medicines and herbal and dietary supplements [including St John's Wort]) that have been taken within 14 days prior to Screening. Drugs that are strong or moderate inhibitors or inducers of cytochrome P450 (CYP)3A4 and/or P-glycoprotein (Pgp) are prohibited
* The use of concomitant medications that prolong the QT/QTc interval
* Study participant has donated more than 500 mL of blood or blood products within 90 days prior to Admission (Day -1) or plans to donate blood during the study (20 weeks post Screening)
* Study participant has consumed any grapefruit, grapefruit juice, grapefruit-containing products, or star fruit within 14 days prior to administration of UCB8600

Part B-specific

* Study participant has:

  1. a history of angioedema, severe asthma, severe food allergies, or anaphylaxis
  2. a personal or family history of cardiomyopathy
* A Screening forced expiratory volume (FEV1) <80% predicted (highest of 3)
* Study participant has:

  1. Allergen immunotherapy, also known as desensitization or hyposensitization at a maintenance licensed dose (depending on the type of immunotherapy [subcutaneous or sublingual]) for ≥3 months prior to Screening and then throughout the study
  2. Severe positive reaction to Screening skin prick test
* Topical or systemic corticosteroids, including high dose oral (>5 mg prednisolone), in the past 14 days prior to Screening and throughout the study
* Topical immunosuppressants in the past 14 days prior to Screening and throughout the study
* Tricyclic antidepressants, prescription antihistamines, over-the-counter antihistamines, and heartburn medications in the past 14 days prior to Admission
* Systemic immunosuppressants such as azathioprine, methotrexate, cyclosporine, and mycophenolate mofetil in the past 4 weeks prior to Screening and throughout the study
* Biologics such as omalizumab for the past 6 months prior to Screening and throughout the study

Part C-specific

* Study participant has:

  1. a history of angioedema, severe asthma, severe food allergies, or anaphylaxis
  2. a personal or family history of cardiomyopathy
* Study participants with a serum IgE level of >1000 kU/L
* A screening FEV1 <80% predicted (average of 3)
* Allergen immunotherapy, also known as desensitization or hyposensitization at a maintenance licensed dose (depending on the type of immunotherapy [subcutaneous or sublingual]) for ≥3 months prior to Screening and then throughout the study
* Topical or systemic corticosteroids, including high dose oral (>5 mg prednisolone), in the past 14 days prior to Screening and throughout the study
* Topical immunosuppressants in the past 14 days prior to Screening and throughout the study
* Systemic immunosuppressants such as azathioprine, methotrexate, cyclosporine, and mycophenolate mofetil in the past 4 weeks prior to Screening and throughout the study
* Biologics such as omalizumab for the past 6 months prior to Screening and throughout the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From Baseline (Day 1) until the End of Study (up to Day 42)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. A treatment-emergent adverse event is characterized according to the intake of the study medication.

SECONDARY OUTCOMES:
The maximum plasma concentration (Cmax) of a single dose UCB8600 | Plasma samples will be taken predose on Day 1 and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, 216 hours postdose
  Cmax: Maximum observed plasma concentration
Time to maximum plasma concentration (tmax) of a single dose UCB8600 | Plasma samples will be taken predose on Day 1 and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, 216 hours postdose
  tmax: Time to maximum observed plasma concentration
The area under the curve (AUC) of a single dose UCB8600 | Plasma samples will be taken predose on Day 1 and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, 216 hours postdose
  AUC0-infinity: Area under the plasma concentration time curve from time 0 to infinity
The maximum plasma concentration (Cmax) of multiple doses UCB8600 | Plasma samples will be taken on Day 1, 9 and 14 at: predose, 0.5, 1, 2, 3, 6, 12, 24 hours postdose
  Cmax: Maximum observed plasma concentration
Time to maximum plasma concentration (tmax) of multiple doses UCB8600 | Plasma samples will be taken on Day 1, 9 and 14 at: predose, 0.5, 1, 2, 3, 6, 12, 24 hours postdose
  tmax: Time to maximum observed plasma concentration
The area under the curve (AUCtau) over a dosing interval on Day 1 of multiple doses UCB8600 | Plasma samples will be taken on Day 1 at: predose, 0.5, 1, 2, 3, 6, 12, 24 hours postdose
  AUCtau: Area Under the Curve over a dosing interval
The area under the curve (AUCtau) over a dosing interval on Day 9 of multiple doses UCB8600 | Plasma samples will be taken on Day 9 at: predose, 0.5, 1, 2, 3, 6, 12, 24 hours postdose
  AUCtau: Area Under the Curve over a dosing interval
The area under the curve (AUCtau) over a dosing interval on Day 14 of multiple doses UCB8600 | Plasma samples will be taken on Day 14 at: predose, 0.5, 1, 2, 3, 6, 12, 24 hours postdose
  AUCtau: Area Under the Curve over a dosing interval

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0086 001, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.